CLINICAL TRIAL: NCT06257875
Title: A Multicenter, Randomized Study to Evaluate the Safety and Efficacy of Lutikizumab for Induction and Maintenance Therapy in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity From Intravenous (IV) and Subcutaneous (SC) Lutikizumab in Adult Participants With Active Ulcerative Colitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M23-703; 2023-505678-14-00 (Other: EU CT)
Record Dates: First submitted 2023-10-02; First posted 2024-02-14 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Lutikizumab; Adalimumab
MeSH Terms: conditions — Colitis, Ulcerative | interventions — lutikizumab; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Induction Group 1 (Experimental): Participants will receive Dose 1 of IV lutikizumab at Baseline followed by SC lutikizumab throughout induction.
  Interventions: Drug: Lutikizumab
- Induction Group 2 (Experimental): Participants will receive Dose 2 of IV lutikizumab at Baseline followed by SC lutikizumab throughout induction.
  Interventions: Drug: Lutikizumab
- Induction Group 3 (Experimental): Participants will receive adalimumab per label throughout induction.
  Interventions: Drug: Adalimumab
- Maintenance Group 1 (Experimental): Participants who responded to lutikizumab induction group 1 or 2 will be re-randomized. Participants in this group will receive SC lutikizumab throughout the maintenance period.
  Interventions: Drug: Lutikizumab
- Maintenance Group 2 (Experimental): Participants who responded to lutikizumab induction group 1 or 2 will be re-randomized. Participants in this group will receive SC lutikizumab throughout the maintenance period.
  Interventions: Drug: Lutikizumab
- Maintenance Adalimumab (Experimental): Participants who respond to adalimumab induction group 3 will continue to receive adalimumab per label in the maintenance period.
  Interventions: Drug: Adalimumab
- Maintenance Non-Responders (Experimental): Participants who do not respond to study drug at the end of induction period will receive SC lutikizumab in the maintenance period.
  Interventions: Drug: Lutikizumab
- Optional Long-Term Extension (LTE) (Experimental): Participants who complete the maintenance period, are willing/able to inject study drug at home, and in whom therapeutic benefit to study drug is confirmed by the investigator, may participate in the optional 52-week LTE.
  Interventions: Drug: Lutikizumab; Drug: Adalimumab

INTERVENTIONS:
Drug: Lutikizumab — Subcutaneous (SC) Injection
  Other Names: ABT-981
  Arms: Induction Group 1; Induction Group 2; Maintenance Group 1; Maintenance Group 2; Maintenance Non-Responders; Optional Long-Term Extension (LTE)
Drug: Lutikizumab — Intravenous (IV) Infusion
  Other Names: ABT-981
  Arms: Induction Group 1; Induction Group 2
Drug: Adalimumab — SC Injection
  Other Names: Humira
  Arms: Induction Group 3; Maintenance Adalimumab; Optional Long-Term Extension (LTE)

SUMMARY:
Ulcerative colitis (UC) is a type of inflammatory bowel disease that causes inflammation and bleeding from the lining of the rectum and colon (large intestine). The purpose of this study is to assess how safe and effective lutikizumab is in adult participants with moderate to severe UC and how lutikizumab compares to adalimumab in the treatment of UC. Adverse events and changes in disease activity will be assessed.

Lutikizumab is an investigational product being developed for the treatment of moderate to severe UC. Participants are placed in groups called treatment arms. Each group receives a different treatment. In the Induction Period, participants will be randomized into 1 of 3 arms receiving lutikizumab Dose 1, lutikizumab Dose 2, or adalimumab. In the Maintenance Period, participants who responded to lutikizumab will be randomized into 1 of 2 arms of lutikizumab maintenance and participants who responded to adalimumab will continue to receive adalimumab. All participants who did not achieve clinical response per modified Mayo Score at the end of the Induction period will receive lutikizumab. Around 200 adult participants with UC will be enrolled at approximately 200 sites worldwide.

During the 12 week Induction Period, participants will be randomized to receive intravenous (IV) and subcutaneous (SC) lutikizumab or SC adalimumab. At the 12 week mark, participants who are on lutikizumab who have responded to treatment will be re-randomized to receive SC lutikizumab at different intervals until Week 52. Participants who are on adalimumab who are responding to treatment will continue to receive adalimumab. Participants who do not respond to treatment will receive SC lutikizumab. Participants who complete the Week 52 visit and in whom therapeutic benefit to study drug is confirmed by the investigator may roll over into an optional, 52-week long-term extension (LTE).

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participant has had a diagnosis of Ulcerative Colitis (UC) for at least 90 days prior to Baseline. Appropriate documentation of biopsy results consistent with the diagnosis of UC in the assessment of the investigator, must be available.
* Active UC with a Modified Mayo Score (mMS) of 5 to 9 points and Mayo Endoscopic Subscore (ESS) of 2 to 3 (confirmed by central review).
* Demonstrated inadequate response to, loss of response to, or intolerance to at least one of the following: oral aminosalicylates, corticosteroids, immunomodulators, and/or advanced therapies.

Exclusion Criteria:

* Current diagnosis of Crohn's Disease (CD) or inflammatory bowel disease-unclassified.
* Extent of inflammatory disease limited to the rectum as assessed by screening endoscopy.
* Prior inadequate response, intolerance or loss of response to adalimumab (including biosimilars). Note: Participant may be enrolled if he/she discontinued adalimumab for reasons other than those listed above (e.g., loss of insurance) or he/she has been exposed to other advanced therapies, including anti-TNFs other than adalimumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-03-23 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Endoscopic Improvement | Week 12
  Endoscopic Improvement is defined as Mayo Endoscopic Subscore (ESS) of 0 or 1. Endoscopies were assessed by a blinded central reader and scored according to the following scale: 0 = Normal appearance of mucosa; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration).
Number of Participants with Adverse Events (AEs) | Up to approximately Week 104
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve Clinical Remission Per Modified Mayo Score (mMS) | Week 12
  Clinical remission on the mMS is defined as Endoscopy subscore = 0 or 1, AND Rectal bleeding subscore = 0, AND Stool frequency subscore <= 1, AND not greater than baseline. The mMS is a composite score of UC disease activity based on the following 3 subscores: SFS, scored from 0 (normal number of stools) to 3 (5 or more stools more than normal); RBS, scored from 0 (no blood seen) to 3 (blood alone passed); ESS, scored from 0 (normal appearance of mucosa) to 3 (severe disease [spontaneous bleeding, ulceration]). The overall mMS ranges from 0 to 9 with higher scores representing more severe disease. The number of responders is calculated based on the total number of participants and estimated response rate, rounding to a nearest whole integer.
Percentage of Participants who Achieve Clinical Response Per mMS | Week 12
  Clinical response per mMS is defined as decrease from baseline >=2 points and >=30%, PLUS a decrease in RBS >= 1 or an absolute RBS <=1. The mMS is a composite score of UC disease activity based on the following 3 subscores: SFS, scored from 0 (normal number of stools) to 3 (5 or more stools more than normal); RBS, scored from 0 (no blood seen) to 3 (blood alone passed); ESS, scored from 0 (normal appearance of mucosa) to 3 (severe disease [spontaneous bleeding, ulceration]). The overall mMS ranges from 0 to 9 with higher scores representing more severe disease. The number of responders is calculated based on the total number of participants and estimated response rate, rounding to a nearest whole integer.
Percentage of Participants who Achieve Endoscopic Remission | Week 12
  Endoscopic remission is defined as Mayo Endoscopic Subscore (ESS) of 0. Endoscopies were assessed by a blinded central reader and scored according to the following scale: 0 = Normal appearance of mucosa; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (191):
- United States (48):
  - Gastro SB /ID# 258331, Chula Vista, California
  - Southern California Res. Ctr. /ID# 258391, Coronado, California
  - Newport Huntington Medical Group /ID# 258371, Huntington Beach, California
  - Om Research LLC /ID# 261383, Lancaster, California
  - UC Irvine Health /ID# 259824, Orange, California
  - University of Colorado Hospital /ID# 258388, Aurora, Colorado
  - Research Associates of South Florida, LLC /ID# 259813, Coral Gables, Florida
  - University of Florida College of Medicine /ID# 260402, Gainesville, Florida
  - Auzmer Research /ID# 260940, Lakeland, Florida
  - Atlantic Medical Research /ID# 258507, Margate, Florida
  - Homestead Associates in Research /ID# 260392, Miami, Florida
  - University of Miami /ID# 258396, Miami, Florida
  - JD Medical Group, LLC /ID# 261235, Miami, Florida
  - Gastroenterology Group Naples /ID# 258346, Naples, Florida
  - AdventHealth Medical Group Blood & Marrow Transplant at Orlando /ID# 260945, Orlando, Florida
  - GCP Clinical Research, LLC /ID# 260401, Tampa, Florida
  - Atlanta Ctr. for Gastro /ID# 259275, Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, LLC /ID# 258359, Macon, Georgia
  - Gastroenterology Consultants, P.C /ID# 258352, Roswell, Georgia
  - Northwestern Medicine - Northwestern Memorial Hospital /ID# 259592, Chicago, Illinois
  - University of Chicago Medical Center /ID# 258491, Chicago, Illinois
  - IU Health University Hospital /ID# 260398, Indianapolis, Indiana
  - Univ Kansas Med Ctr /ID# 258489, Kansas City, Kansas
  - Louisiana Research Center, LLC /ID# 258330, Shreveport, Louisiana
  - Massachusetts General Hospital /Id# 259817, Boston, Massachusetts
  - Clin Res Inst of Michigan, LLC /ID# 258386, Chesterfield, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 259267, Chesterfield, Michigan
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinic /ID# 258493, Wyoming, Michigan
  - Mayo Clinic - Rochester /ID# 258402, Rochester, Minnesota
  - Univ New Mexico /ID# 258490, Albuquerque, New Mexico
  - NY Scientific /ID# 260937, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Associates /ID# 258504, Lake Success, New York
  - Weill Cornell Medicine/NYP /ID# 258953, New York, New York
  - Columbia University Medical Center /ID# 258496, New York, New York
  - Atrium Health /ID# 258506, Charlotte, North Carolina
  - DJL Clinical Research, PLLC /ID# 259465, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 260387, Winston-Salem, North Carolina
  - Plains Clinical Research Center, LLC /ID# 258502, Fargo, North Dakota
  - Digestive Disease Specialists /ID# 258499, Oklahoma City, Oklahoma
  - Digestive Health Associates of Texas (DHAT) Research Institute - Garland /ID# 258358, Garland, Texas
  - Baylor College of Medicine /ID# 258394, Houston, Texas
  - BioStar Clinical Research Group - Houston - Katy Freeway /ID# 261164, Houston, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 258403, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 258347, San Antonio, Texas
  - Tyler Research Institute, LLC /ID# 258383, Tyler, Texas
  - Texas Digestive Disease Consultants - Webster /ID# 258718, Webster, Texas
  - University Physicians and Surgeons Inc. /ID# 260399, Huntington, West Virginia
  - Wisconsin Center for Advanced Research /ID# 258949, Milwaukee, Wisconsin
- Australia (5):
  - Bankstown-Lidcombe Hospital /ID# 259089, Bankstown, New South Wales
  - Lyell McEwin Hospital /ID# 260580, Elizabeth Vale, South Australia
  - The Queen Elizabeth Hospital /ID# 259482, Woodville South, South Australia
  - St Vincent's Hospital Melbourne /ID# 259473, Fitzroy Melbourne, Victoria
  - Fiona Stanley Hospital /ID# 259480, Murdoch, Western Australia
- Austria (2):
  - Universitaetsklinikum St. Poelten /ID# 258256, Sankt Pölten, Lower Austria
  - Medizinische Universitaet Wien /ID# 258026, Vienna, Vienna
- Belgium (6):
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 258214, Anderlecht, Brussels Capital
  - UZ Gent /ID# 258210, Ghent, Oost-Vlaanderen
  - Vitaz /Id# 258222, Sint-Niklaas, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 258226, Leuven, Vlaams-Brabant
  - AZ Maria Middelares /ID# 258219, Ghent
  - CHU de Liege /ID# 258212, Liège
- Bulgaria (7):
  - Hospital Tsaritsa Yoanna /ID# 258338, Sofiya, Sofia
  - Medical Center - Doverie /ID# 261936, Sofiya, Sofia
  - ACIBADEM City Clinic Diagnostic-Consultative Center /ID# 258339, Sofiya, Sofia
  - Umbal Kaspela /ID# 258336, Plovdiv
  - 2nd Mhat /ID# 258337, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 261417, Sofia
  - UMHAT Multiprofile Hospital for Active Treatment Sveta Marina /ID# 258878, Varna
- Canada (3):
  - Gastroenterology and Internal Medicine Research Institution /ID# 258765, Edmonton, Alberta
  - Covenant Health /ID# 258799, Edmonton, Alberta
  - Toronto Digestive Disease Associates /ID# 260460, Vaughan, Ontario
- Croatia (5):
  - Klinicki bolnicki centar Zagreb /ID# 258145, Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 258147, Zagreb, City of Zagreb
  - POLIKLINIKA BORZAN d.o.o. /ID# 258146, Osijek, County of Osijek-Baranja
  - Specialty Hospital Medico /ID# 258169, Rijeka, Primorje-Gorski Kotar County
  - Klinicki Bolnicki Centar (KBC) Split /ID# 258153, Split, Split-Dalmatia County
- Estonia (4):
  - West Tallinn Central Hospital /ID# 262035, Tallinn, Harju
  - Medicum /ID# 268320, Tallinn, Harju
  - Parnu Hospital /ID# 261783, Pärnu
  - Tartu University Hospital /ID# 261782, Tartu
- France (5):
  - Chu de Nice-Hopital L'Archet Ii /Id# 258041, Nice, Alpes-Maritimes
  - CHU Toulouse - Hopital Rangueil /ID# 258044, Toulouse, Haute-Garonne
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 258555, Créteil, Paris
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 258042, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord /ID# 258040, St-Priest-en-Jarez, Pays de la Loire Region
- Germany (6):
  - Universitaetsklinikum Ulm /ID# 258616, Ulm, Baden-Wurttemberg
  - Klinikum rechts der Isar /ID# 260228, Munich, Bavaria
  - St. Marien- und St. Annastiftskrankenhaus /ID# 264691, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Eugastro /ID# 260229, Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 258614, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 258617, Hamburg
- Greece (4):
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 257831, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 257832, Heraklion, Crete
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 257829, Athens
  - General Hospital of Thessaloniki Hippokrateio /ID# 260810, Thessaloniki
- Hungary (5):
  - Clinfan /ID# 258094, Szekszárd, Tolna County
  - Clinexpert Kft /ID# 258449, Budapest
  - Synexus Hungary Clinical Research Centre - Budapest /ID# 258915, Budapest
  - Semmelweis Egyetem /ID# 258527, Budapest
  - Szegedi Tudományegyetem /ID# 258095, Szeged
- Ireland (2):
  - St Vincents University Hospital /ID# 261560, Elm Park, Dublin
  - Beaumont Hospital /ID# 261561, Dublin
- Israel (6):
  - Yitzhak Shamir Medical Center /ID# 258533, Ẕerifin, Central District
  - Shaare Zedek Medical Center /ID# 258529, Jerusalem, Jerusalem
  - Soroka University Medical Center /ID# 258530, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 258532, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 258528, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 258531, Petah Tikva
- Italy (4):
  - Azienda Ospedaliero Universitaria di Cagliari - P.O. Duilio Casula /ID# 258455, Monserrato, Cagliari
  - Azienda Ospedaliera San Camillo Forlanini /ID# 258453, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 258452, Rome, Roma
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 258456, Negrar, Verona
- Japan (24):
  - Gamagori City Hospital /ID# 260682, Gamagori-shi, Aichi-ken
  - Aichi Medical University Hospital /ID# 258867, Nagakute, Aichi-ken
  - Tsujinaka Hospital - Kashiwanoha /ID# 258548, Kashiwa-shi, Chiba
  - Juntendo University Urayasu Hospital /ID# 259582, Urayasu-shi, Chiba
  - Kitakyushu Municipal Medical Center /ID# 259600, Kitakyushu-shi, Fukuoka
  - Fukushima Medical University Hospital /ID# 259591, Fukushima, Fukushima
  - Gifu University Hospital /ID# 259572, Gifu, Gifu
  - Ogaki Municipal Hospital /ID# 259905, Ogaki-shi, Gifu
  - National Hospital Organization Fukuyama Medical Center /ID# 258861, Fukuyama-shi, Hiroshima
  - Aoyama Clinic /ID# 259587, Kobe, Hyōgo
  - Hyogo Medical University Hospital /ID# 258827, Nishinomiya-shi, Hyōgo
  - Sameshima Hospital /ID# 259589, Kagoshima, Kagoshima-ken
  - Kagoshima IBD Gastroenterology Clinic /ID# 259603, Kagoshima, Kagoshima-ken
  - Sai Gastroenterology and Proctology Clinic /ID# 260832, Fujidera-shi, Osaka
  - Kinshukai Infusion Clinic /ID# 259588, Osaka, Osaka
  - Saga University Hospital /ID# 259625, Saga, Saga-ken
  - Tokitokai Tokito clinic /ID# 259036, Saitama-shi, Saitama
  - Hamamatsu University Hospital /ID# 259580, Hamamatsu, Shizuoka
  - NHO Shizuoka Medical Center /ID# 259033, Sunto-gun, Shizuoka
  - Institute of Science Tokyo Hospital /ID# 259003, Bunkyo-ku, Tokyo
  - Tokai University Hachioji Hospital /ID# 258897, Hachioji-shi, Tokyo
  - Kyorin University Hospital /ID# 259843, Mitaka-shi, Tokyo
  - Center hospital of the National Center for Global Health and Medicine /ID# 259598, Shinjuku-ku, Tokyo
  - Toyama Prefectural Central Hospital /ID# 259499, Toyama, Toyama
- Latvia (3):
  - SIA Polana-D /ID# 262932, Daugavpils
  - Liepaja Regional Hospital /ID# 261484, Liepāja
  - Pauls Stradins Clinical University Hospital /ID# 261483, Riga
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 261486, Kaunas
  - Panevezys Republican Hospital /ID# 261780, Panevezys
  - Vilnius University Hospital Santaros Klinikos /ID# 261487, Vilnius
- New Zealand (3):
  - Dunedin Hospital /ID# 258584, Otago, Otago
  - Waikato Hospital /ID# 258607, Hamilton, Waikato Region
  - Hutt Hospital /ID# 258608, Lower Hutt, Wellington Region
- Norway (2):
  - Akershus Universitetssykehus /ID# 261586, Nordbyhagen, Akershus
  - Universitetssykehuset I Nord-Norge /ID# 261649, Tromsø, Troms
- Poland (7):
  - Gastromed Sp. z o.o /ID# 258310, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Melita Medical /ID# 258379, Wroclaw, Lower Silesian Voivodeship
  - Medrise Sp. z o.o. /ID# 258561, Lublin, Lublin Voivodeship
  - Centrum Medyczne Lukamed Sp. z o.o. /ID# 258457, Chojnice, Pomeranian Voivodeship
  - H-T Centrum Medyczne Endoterapia /ID# 258540, Tychy, Silesian Voivodeship
  - Twoja Przychodnia SCM /ID# 259280, Szczecin, West Pomeranian Voivodeship
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Sp. j. /ID# 258842, Ksawerów, Łódź Voivodeship
- Puerto Rico (3):
  - Clinical Research Investigator Group, LLC /ID# 260647, Bayamón
  - Caribbean Medical Research Center /ID# 268395, San Juan
  - School of Medicine University of Puerto Rico-Medical Science Campus /ID# 258508, San Juan
- Serbia (6):
  - Clinical Hosp Center Zvezdara /ID# 257766, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 257764, Belgrade, Beograd
  - Clinical Hospital Center Dr Dragisa Misovic - Dedinje /ID# 257768, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 257765, Belgrade, Beograd
  - General Hospital Leskovac /ID# 257767, Leskovac, Jablanicki Okrug
  - University Clinical Center Vojvodina /ID# 257763, Novi Sad
- Slovenia (3):
  - General Hospital Celje /ID# 261482, Celje
  - Univ Medical Ctr Ljubljana /ID# 261474, Ljubljana
  - Splosna bolnisnica Murska Sobota /ID# 262486, Murska Sobota
- South Africa (4):
  - Clinresco Centers /ID# 258431, Johannesburg, Gauteng
  - Johese Clinical Research Midstream /ID# 260195, Pretoria, Gauteng
  - Private Practice Dr MN Rajabally /ID# 260671, Cape Town, Western Cape
  - Spoke Research Inc /ID# 258432, CAPE TOWN Milnerton, Western Cape
- South Korea (6):
  - Inje University Haeundae Hospital /ID# 258822, Busan, Busan Gwang Yeogsi
  - Dong-A University Medical Center /ID# 258423, Busan, Busan Gwang Yeogsi
  - The Catholic University of Korea, Daejeon St. Mary's Hospital /ID# 258424, Daejeon, Daejeon Gwang Yeogsi
  - Kangbuk Samsung Hospital /ID# 258416, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 258420, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 258422, Seoul
- Spain (4):
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 259114, Santiago de Compostela, A Coruna
  - Hospital Universitario de Navarra /ID# 258173, Pamplona, Navarre
  - Hospital Universitario La Paz /ID# 258172, Madrid
  - Hospital Universitario Virgen Macarena /ID# 258175, Seville
- Switzerland (2):
  - Inselspital, Universitaetsspital Bern /ID# 260106, Bern
  - Intesto /ID# 260114, Bern
- Taiwan (4):
  - National Taiwan University Hospital /ID# 258476, Taipei City, Taipei
  - National Taiwan University Hospital - Hsinchu branch /ID# 259422, Hsinchu
  - China Medical University Hospital /ID# 258478, Taichung
  - Linkou Chang Gung Memorial Hospital /ID# 258724, Taoyuan
- United Kingdom (5):
  - Addenbrookes Hospital /ID# 258744, Cambridge, Cambridgeshire
  - Gartnavel General Hospital /ID# 258741, Glasgow, Glasgow City
  - Dup_Guys and St Thomas NHS Foundation Trust - Guy's Hospital /ID# 258730, London, Greater London
  - Oxford University Hospitals NHS Foundation Trust /ID# 258745, Oxford, Oxfordshire
  - Barts Health NHS Trust /ID# 258600, London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-703